CLINICAL TRIAL: NCT02037087
Title: The Impact of Prenatal Short Messages on Maternal and Newborn Health
Brief Title: The Impact of Prenatal Short Messages (SMS) on Maternal and Newborn Health
Acronym: SMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Yanfang Su, ScD, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Factorial | Masking: Single
Other Study IDs: newborn2013
Record Dates: First submitted 2014-01-14; First posted 2014-01-15 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Short Message Service; Text Messaging
Keywords: Short Message Service; newborn health; maternal behavior; good household pregnancy practice; care seeking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Good household prenatal practice (GHPP) (Experimental): The GHPP arm receives SMS messages regarding knowledge on nutrition, labor, non-medical pain management, breastfeeding, and depression. This arm also receives messages delivered to the control group.
  Interventions: Behavioral: Good household prenatal practice
- Care seeking (CS) (Experimental): The CS arm receives SMS messages which include danger-sign recognition and reminders for government-subsidized projects. This arm also receives messages delivered to the control group.
  Interventions: Behavioral: Care seeking
- Full bank of SMS (Experimental): This arm receives the SMS messages delivered to the GHPP, CS and control group.
  Interventions: Behavioral: Full bank of SMS
- Control (No Intervention): Control group receives SMS messages regarding:
  * Reminders of prenatal visits and certified skilled attendance of labor (status quo);
  * Fetal development in different gestational stages.
  The three experimental groups receive the control messages as well.

INTERVENTIONS:
Behavioral: Good household prenatal practice — Knowledge on nutrition, labor, non-medical pain management, breastfeeding and depression
  Arms: Good household prenatal practice (GHPP)
Behavioral: Care seeking — * Danger-sign recognition
  * Reminders for government projects
  Arms: Care seeking (CS)
Behavioral: Full bank of SMS — * Danger-sign recognition
  * Reminders for government projects
  * Knowledge on nutrition, labor, non-medical pain management, breastfeeding and depression
  Arms: Full bank of SMS

SUMMARY:
It is hypothesized that delivering short messages (SMS) to pregnant women can improve maternal and newborn health outcomes. This pilot offers mothers-to-be in rural China free daily short messages (SMS) via cell phone. The aim is to advise them on (a) good household prenatal practices (GHPP) and (b) care seeking (CS) in order to improve the quality of life for mothers and newborns.

DETAILED DESCRIPTION:
Factorial quasi-randomization is utilized to compare two groups of interventions (i.e., GHPP and CS) as well as to compare these individual interventions with a combination of the interventions. It is also possible that distinct treatments have interaction effects, and we plan to test for this. Policymakers are interested in using different strategies to enhance neonatal health. For example, the bank of SMS developed by our team is a combination of several components: reminders for regular checkups, information on GHPP, and information on CS. From a policy perspective, the evaluation of the full bank of SMS may be sufficient for the government to decide whether or not to scale up the full bank of SMS. However, to understand maternal behavior and, for policy purposes, to understand which components in the bank of SMS should be scaled up, it is important to disentangle which component contributes most to final neonatal health. Taken together, are all the components of the bank of SMS effective in changing maternal behavior and enhancing neonatal health? Which mechanisms are at play, good household prenatal care, care seeking in pregnancy, or both?

ELIGIBILITY:
There were two inclusion criteria: Local pregnant women must 1) own a cell phone in the household, and 2) visit a MCHC for antenatal care during pregnancy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4467 (Actual)
Dates: Start 2013-09; Primary Completion 2015-10 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Newborn health | the first month after birth
  Newborn health is measured by appropriateness of weight for gestational age.

SECONDARY OUTCOMES:
Neonatal Adverse Outcome Indicator (NAOI) | the first month after birth
  The NAOI focuses on measuring severe neonatal morbidity.
Actual number of prenatal visits over expected visits | In the duration of pregnancy, an expected average of 9 months
Uptake of government-subsidized programs | In the duration of pregnancy, an expected average of 9 months, and 1 month after birth
  This outcome is measured by the following metrics:
  1. Duration of folic acid
  2. Uptake of infant vaccinations
C-section rate | child birth
Maternal health | Child birth and 1 year after birth
  Maternal health is measured by change of perception in general health and postpartum depression.
Near-miss | In the duration of pregnancy, an expected average of 9 months, and childbirth
  The near-miss focuses on measuring severe maternal morbidity.
Psychological outcomes | In the duration of pregnancy, an expected average of 9 months
  Attitudes, personal norms, self-efficacy, social desirability, intentions, plans, susceptibility, expectations, and severity

CONTACTS AND LOCATIONS:
Overall Officials: Yanfang Su, MA, Principal Investigator — Harvard School of Public Health (HSPH); Zhongliang Zhou, PhD, Principal Investigator — Xi'an Jiaotong University; Changzheng Yuan, MS, Principal Investigator — Harvard School of Public Health (HSPH); Jesse Heitner, MPP, Principal Investigator — Harvard School of Public Health (HSPH); Benjamin Campbell, BA, Principal Investigator — Dartmouth College
Locations (1):
- Xi'an Jiaotong University, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Su Y, Heitner J, Yuan C, Si Y, Wang D, Zhou Z, Zhou Z. Effect of a Text Messaging-Based Educational Intervention on Cesarean Section Rates Among Pregnant Women in China: Quasirandomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Nov 3;8(11):e19953. doi: 10.2196/19953. PMID 33141099
- [Derived] Su Y, Yuan C, Zhou Z, Heitner J, Campbell B. Impact of an SMS advice programme on maternal and newborn health in rural China: study protocol for a quasi-randomised controlled trial. BMJ Open. 2016 Aug 10;6(8):e011016. doi: 10.1136/bmjopen-2015-011016. PMID 27515750